CLINICAL TRIAL: NCT03104075
Title: Genomics and Epigenomics of the Elderly Response to Pneumococcal Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Jackson Laboratory (Other)
Collaborators: UConn Health (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-071J-1
Record Dates: First submitted 2017-03-21; First posted 2017-04-07 (Actual); Results first posted 2021-12-07 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pneumonia; Aging
Keywords: Genomics; Epigenomics; Pneumococcal vaccine; Elderly
MeSH Terms: conditions — Pneumonia | interventions — 13-valent pneumococcal vaccine; Pneumococcal Vaccines; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Intervention Model Description: Randomized assignment to group will be in a 1:1 ratio utilizing block randomization in blocks of 10 to receive Prevnar-13 or Pneumovax 23. Following randomized assignment of vaccine, the study will be open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prevnar 13 (Active Comparator): Prevnar 13 (Pneumococcal 13valent Conj Vaccine Diphtheria CRM197 Protein) will be administered at the single 0.5 ml dose, by intramuscular injection with routine clinical care.
  Interventions: Biological: Pneumococcal 13valent Conj Vaccine Diphtheria CRM197 Protein
- Pneumovax 23 (Active Comparator): Pneumovax 23 (Pneumococcal Vaccine Polyvalent) will be administered at the single 0.5ml dose, by intramuscular injection with routine clinical care.
  Interventions: Biological: Pneumococcal Vaccine Polyvalent

INTERVENTIONS:
Biological: Pneumococcal 13valent Conj Vaccine Diphtheria CRM197 Protein — One to two years after receiving the randomly-assigned vaccination, participants may opt to receive administration of a second pneumococcal vaccine with Pneumovax 23
  Other Names: Prevnar 13
  Arms: Prevnar 13
Biological: Pneumococcal Vaccine Polyvalent — One to two years after receiving the randomly-assigned vaccination, participants may opt to receive administration of a second pneumococcal vaccine with Prevnar-13
  Other Names: Pneumovax 23
  Arms: Pneumovax 23

SUMMARY:
This is a prospective, single-site, randomized, then open-label study designed to develop a detailed transcriptional and epigenetic profile of the immune response to pneumococcal vaccination with conjugated and non-conjugated polysaccharide vaccines in the senescent immune system of older adults.

In this study, 40 healthy adults ages 60 and older that have never received pneumococcal vaccination, will be randomized in a 1:1 ratio to receive Prevnar-13 (Pfizer), a conjugated 13-valent vaccine or Pneumovax 23 (Merck), a non-conjugated 23-valent vaccine. Following randomized assignment of vaccine, the study will be open-label.

Six (6) study visits will occur over about 70 days, with an optional 7th visit for participants to receive a second vaccination with the other pneumococcal vaccine one to two years after randomization. Participants will provide blood samples for transcriptional, epigenetic and biological analyses pre- and post-vaccination.

DETAILED DESCRIPTION:
This prospective, single-site, randomized, then open-label study is designed to develop a detailed transcriptional and epigenetic profile of the immune response to pneumococcal vaccination with conjugated and non-conjugated polysaccharide vaccines in the senescent immune system of older adults. This knowledge may lead to development of more effective vaccines through increased understanding of the effects of immunosenescence on mechanisms of immune response to pneumococcal vaccination in older adults elderly.

Forty (40) healthy adults ages 60 and older that have never received pneumococcal vaccination, will be randomized in a 1:1 ratio to receive Prevnar-13 (Pfizer), a conjugated 13-valent vaccine or Pneumovax 23 (Merck), a non-conjugated 23-valent vaccine. Following randomized assignment of vaccine, the study will be open-label. The study sample will be drawn from the population of healthy older participants in the catchment area of UConn Health in Farmington, CT.

The first six (6) study visits are planned to occur over 67 days at Days -7, 0, 1, 10, 28 (±3 d) and 60 (± 5d). Participants will provide blood samples for transcriptional, epigenetic and biological analyses pre- and post-vaccination.

One to two years after receiving the randomly-assigned vaccination, participants may opt to receive administration of a second pneumococcal vaccine with the vaccine that they did not receive by random assignment at Visit 2 (Day 0). This second vaccine will be provided at no charge to the participant. Administration of this vaccine will occur at an optional Visit 7 for participants who choose to receive the second vaccine and will be scheduled at the participant's convenience one-two years after receiving the first pneumococcal vaccine.

If the participant opts to receive the second vaccine within the study and attends optional Visit 7, blood samples for genomic and biologic analysis will be collected at the visit.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent
* Male or Female, 60 years of age or older
* Willing to receive pneumococcal vaccination with Prevnar 13 (Wyeth/ Pfizer) or Pneumovax 23 (Merck), as randomly assigned.
* Available to attend 6 study visits over 67 days (Visit 7 is optional at Day 365-720).

Exclusion Criteria:

* Previous pneumococcal vaccination with Prevnar 13 or Pneumovax 23.
* History of anaphylactic/anaphylactoid or severe allergic reaction to any component of Pneumovax 23, Prevnar 13 or any diphtheria toxoid-containing vaccine.
* Established diagnosis of diabetes
* History of receiving Zostavax (shingles vaccine) within previous 4 weeks. (Study entry may be delayed to satisfy a 28-day interval between vaccinations)
* Known history of any of the following co-morbid conditions:

  * Malignancy (participants without a recurrence in the last 5 years will be allowed)
  * Congestive Heart Failure
  * Cardiovascular Disease (unstable ≤ 6 months*)
  * Kidney disease
  * Renal failure
  * Impaired hepatic function
  * Autoimmune disease such as: Rheumatoid Arthritis, systemic lupus erythematosus (SLE), Inflammatory Bowel Disease, etc.
  * Use of medicines during past 6 months known to alter immune response such as high-dose corticosteroids
  * HIV, AIDS or other Immunodeficiency
  * Recent (≤ 3 months) trauma or surgery
  * Current substance and/or alcohol abuse * Unstable disease is defined as a change in therapy or hospitalization for worsening disease.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Kuchel, M.D. F.R.C.P, Principal Investigator — UConn Center on Aging
Locations (1):
- UConn Center On Aging, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants will provide or decline consent within the ICF for sharing of their randomly recoded (new code that is different than the study code) genomic data in public and/or controlled access scientific databases. The study database will include a field for whether consent for genomic data sharing was provided or declined by the participant and if consent provided was for public and/or limited access databases. This information will be included in the dataset so that it can be provided to dbGAP (NIH database of Genotypes and Phenotypes) at the conclusion of the study to ensure that the wishes of the participant regarding use of their data and samples are respected.
  Raw IPD data is available through dbGAP (phs002361) due to patient privacy concerns.
  Genomic summary results and gene expression data are shared on GEO; accession numbers GSE247276 (Bulk) and GSE247277 (scRANSeq).
Time Frame: Conclusion of study
Access Criteria: GEO open access Raw IPD controlled-access dbGaP per accession number above.

REFERENCES:
- [Background] Thibodeau A, Eroglu A, McGinnis CS, Lawlor N, Nehar-Belaid D, Kursawe R, Marches R, Conrad DN, Kuchel GA, Gartner ZJ, Banchereau J, Stitzel ML, Cicek AE, Ucar D. AMULET: a novel read count-based method for effective multiplet detection from single nucleus ATAC-seq data. Genome Biol. 2021 Sep 1;22(1):252. doi: 10.1186/s13059-021-02469-x. PMID 34465366
- [Result] Ravichandran S, Erra-Diaz F, Karakaslar OE, Marches R, Kenyon-Pesce L, Rossi R, Chaussabel D, Pascual V, Palucka K, Paust S, Nahm MH, Kuchel GA, Banchereau J, Ucar D. Distinct baseline immune characteristics associated with responses to conjugated and unconjugated pneumococcal polysaccharide vaccines in older adults. medRxiv [Preprint]. 2023 Apr 19:2023.04.16.23288531. doi: 10.1101/2023.04.16.23288531. PMID 37131707

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevnar 13 | Pneumovax 23
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Participant did not complete the last study visit due to hospitalization unrelated to the vaccine | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant was not included in the baseline data analysis because their blood serum samples were not collected. As a result, the researchers were not able to calculate the baseline OPA titers for this participant to include them in further data analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prevnar 13 | Pneumovax 23 | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.52 (7.15) | 69.25 (9.25) | 68.40 (7.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.83 (3.77) | 27.16 (5.94) | 26.13 (5.04)

OUTCOME MEASURES:

1. Primary Outcome: Pneumococcal-specific Antibody Responses
Description: To vaccinate healthy older participants with pneumococcal vaccines, collect longitudinal blood samples and assess pneumococcal-specific antibody responses. The unit of measurement used is log2 titer defined as a measure to quantify the overall strength of responses using the sum of all serotype responses. Data shown below is from longitudinal study timepoints (pre and post) first pneumococcal vaccine. At study endpoint, Visit 7, a second pneumococcal vaccine was administered and no further sample collection visits were conducted as proposed in the study design.
Time Frame: 70 days
Population: 39 healthy volunteers
Measure: Mean (Standard Deviation); unit: log2 titer
Groups:
- Prevnar 13: Prevnar 13 (Pneumococcal 13valent Conj Vaccine Diphtheria CRM197 Protein) will be administered at the single 0.5 ml dose, by intramuscular injection with routine clinical care. [Data analyzed and shown below for the first vaccine i.e. Prevnar 13]
  Pneumococcal 13valent Conj Vaccine Diphtheria CRM197 Protein: One to two years after receiving the randomly-assigned vaccination, participants may opt to receive administration of a second pneumococcal vaccine with Pneumovax 23. [Second vaccine i.e. Pneumovax 23 administered at study endpoint (Visit 7), no further data collected post-second vaccination]
- Pneumovax 23: Pneumovax 23 (Pneumococcal Vaccine Polyvalent) will be administered at the single 0.5ml dose, by intramuscular injection with routine clinical care. [Data analyzed and shown below for the first vaccine i.e. Pneumovax 23]
  Pneumococcal Vaccine Polyvalent: One to two years after receiving the randomly-assigned vaccination, participants may opt to receive administration of a second pneumococcal vaccine with Prevnar-13. [Second vaccine i.e. Prevnar 13 administered at study endpoint (Visit 7), no further data collected post-second vaccination]
Arm/Group | Prevnar 13 | Pneumovax 23
Number analyzed (Participants) | 19 | 20
log2 titer
  Baseline | 72.1 (19.4) | 79.4 (18.6)
  Post first vaccination | 128.9 (19.5) | 120.9 (15.0)

2. Primary Outcome: Pneumococcal-specific Antibody Responses - Fold Change Post First Vaccination
Description: Fold change between the baseline and post first vaccination titers was calculated for each pneumococcal vaccine cohort.
  Data shown below is from longitudinal study timepoints (pre and post) first pneumococcal vaccine. At study endpoint, Visit 7, a second pneumococcal vaccine was administered and no further sample collection visits were conducted as proposed in the study design.
Time Frame: 70 days
Population: 39 healthy volunteers
Measure: Mean (Standard Deviation); unit: Fold Change
Arm/Group | Prevnar 13 | Pneumovax 23
Number analyzed (Participants) | 19 | 20
Fold Change | 55.6 (25.5) | 41.6 (18.8)

3. Secondary Outcome: Number of Genes Upregulated Following Vaccination With PCV13 or PPSV23
Description: RNA-seq and ATAC-seq to enable quantitative assessment of both coding RNA's and ncsRNA's as well as to resolve the epigenetic landscape of immune cells in the context of vaccine responses. We assessed the number of genes upregulated post first vaccination [PCV13 or PPSV23].
  Data shown below is from longitudinal study timepoints (pre and post) first pneumococcal vaccine. At study endpoint, Visit 7, a second pneumococcal vaccine was administered and no further sample collection visits were conducted as proposed in the study design.
Time Frame: 10 days post first vaccination
Population: To compare the transcriptional responses induced by vaccines on circulating PBMCs we generated RNA-seq data from 31 responders out of 39 total donors. We selected the topmost strong and weak responders from each participant arm (15 participants in Prevnar 13 arm, 16 participants in Pneumovax 23 arm) to generate RNA-seq data. The aim was to identify specific RNA transcriptional signatures of responsivity vs non-responsivity to the first administered pneumococcal vaccine.
Measure: Number; unit: Number of upregulated genes at day 10
Arm/Group | Prevnar 13 | Pneumovax 23
Number analyzed (Participants) | 15 | 16
Number of upregulated genes at day 10 | 26 | 42

4. Secondary Outcome: Alterations to APCs, Tfh Cells or B Cells in Response to PCV13 and PPSV23
Description: Measure of functional status of immune cells in older participants following administration of a single pneumococcal vaccine, Prevnar13 or Pneumovax23, at baseline and 10 days post first vaccination.
  Data shown below is from longitudinal study timepoints (pre and post) first pneumococcal vaccine. At study endpoint, Visit 7, a second pneumococcal vaccine was administered and no further sample collection visits were conducted as proposed in the study design.
Time Frame: baseline and 10 days post first vaccination
Population: A longitudinal analysis of different cell populations in whole blood samples was performed using flow cytometry at various time points. The number of plasmablasts and ICOS+ Tfh cells at baseline and post first vaccination at day 10 are reported below.
Measure: Mean (Standard Deviation); unit: cells/microliter
Arm/Group | Prevnar 13 | Pneumovax 23
Number analyzed (Participants) | 19 | 20
cells/microliter
  Plasmablasts cell count at baseline | 0.4 (0.4) | 0.5 (0.3)
  Plasmablasts cell count at Day 10 post first vaccination | 0.7 (0.8) | 1.6 (2.5)
  ICOS+Tfh cell count at baseline | 4.1 (3.8) | 4.1 (2.4)
  ICOS+Tfh cell count at Day 10 post first vaccination | 8.8 (7.6) | 6.8 (3.9)

ADVERSE EVENTS:
Time Frame: Data were collected on participants during the 2017-2018 vaccination seasons. Blood samples obtained 7 days prior to vaccination and Day 1, 10, 28, 60 post-vaccination.
Description: AEs were collected on participants throughout the duration of the study. None of the AEs were related to the vaccine. One participant had a vasovagal syncope episode due to blood draw.
Arm/Group | Prevnar 13 | Pneumovax 23
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 1/19 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevnar 13 (N=19) | Pneumovax 23 (N=20)
Vasovagal Syncope (General disorders) | 1 (1) | 0 (0) — Vasovagal episode due to blood draw

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT03104075/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT03104075/ICF_001.pdf